CLINICAL TRIAL: NCT02664220
Title: A Randomized Pilot Trial of Dilute Povidone-iodine Irrigation vs No Irrigation for Children With Acute, Perforated Appendicitis
Brief Title: Dilute Povidone-iodine Irrigation vs No Irrigation for Children With Acute, Perforated Appendicitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, KuoJen Tsao, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-15-1000
Record Dates: First submitted 2015-12-21; First posted 2016-01-26 (Estimated); Results first posted 2019-04-17 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-03

CONDITIONS: Acute, Perforated Appendicitis
Keywords: Povidone-iodine irrigation
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Povidone-iodine irrigation (Experimental)
  Interventions: Drug: Povidone-iodine irrigation
- No irrigation (Active Comparator)
  Interventions: Procedure: No irrigation

INTERVENTIONS:
Drug: Povidone-iodine irrigation — Povidone-iodine (PVI) is an antiseptic solution consisting of polyvinylpyrrolidone with water, iodide, and 1% available iodine. It has bactericidal ability against a large array of pathogens, including those pathogens which commonly cause postoperative IAA in children with perforated appendicitis.
  1% PVI will be used. Once the appendix has been removed and hemostasis ensured, the surgeon will perform the irrigation with 10cc/kg (minimum 100ml and maximum 1000ml) of 1% PVI. After completing the irrigation, the surgeon will suction out all intra-abdominal fluid into a suction canister.
  Arms: Povidone-iodine irrigation
Procedure: No irrigation — Patients allocated to the control group will not undergo intra-abdominal irrigation.
  Arms: No irrigation

SUMMARY:
The goal of this study is to compare the efficacy of PVI irrigation to no irrigation for decreasing postoperative intra-abdominal abscesses in children with perforated appendicitis. Additionally, this study aims to verify the safety profile of dilute PVI for intra-abdominal irrigation.

DETAILED DESCRIPTION:
Postoperative intra-abdominal abscesses are common occurrences after perforated appendicitis in pediatric patients despite utilization of evidence-based practices. Povidone-iodine is a commonly used antiseptic in surgical procedures and has been shown to be effective in reducing postoperative abscesses in adults with perforated appendicitis. This trial will be the first to rigorously test the efficacy of povidone-iodine irrigation in children and to verify its safety profile in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Children who undergo an appendectomy for perforated appendicitis. (Appendicitis: Diagnosis is made intraoperatively by the surgeon. Diagnosis Method: The visualization of a gross defect in the appendiceal wall or the presence of intraperitoneal stool or a fecalith at the time of operation.)

Exclusion Criteria:

* Patients presenting with simple or gangrenous appendicitis
* Patients with a history of iodine sensitivity, thyroid disease or renal disease
* Patients undergoing interval or incidental appendectomy
* Patients/parents/legal guardians who are both non-English and non-Spanish speaking

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2016-04; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: KuoJen Tsao, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

REFERENCES:
- [Derived] Anderson KT, Putnam LR, Bartz-Kurycki MA, Hamilton EC, Yafi M, Pedroza C, Austin MT, Kawaguchi AL, Kao LS, Lally KP, Tsao K. Povidone-iodine Irrigation for Pediatric Perforated Appendicitis May Be Protective: A Bayesian Pilot Randomized Controlled Trial. Ann Surg. 2020 May;271(5):827-833. doi: 10.1097/SLA.0000000000003398. PMID 31567357

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 372 subjects consented, 100 were enrolled as these subjects had perforated appendicities
Period: Overall Study
Arm/Group | Povidone-iodine Irrigation | No Irrigation
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Povidone-iodine Irrigation | No Irrigation | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 50 | 50 | 100
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.4 (3.6) | 10.6 (4) | 10.4 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 22 | 40
  Male | 32 | 28 | 60
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 8 | 11 | 19
  Hispanic | 29 | 28 | 57
  Black | 5 | 4 | 9
  Asian | 2 | 0 | 2
  Other/Unknown | 6 | 7 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Postoperative Intra-abdominal Abscess
Description: 30 days postoperative intra-abdominal abscess was confirmed by an image using a standardized definition and protocol
Time Frame: 30 days post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Povidone-iodine Irrigation | No Irrigation
Number analyzed (Participants) | 50 | 50
Participants | 6 | 8

2. Secondary Outcome: Total Hospital Length of Stay
Description: Total hospital length of stay will be the aggregate of all days in the hospital including any appendicitis-related readmissions within 30 postoperative days.
Time Frame: 30 days post surgery
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Povidone-iodine Irrigation | No Irrigation
Number analyzed (Participants) | 50 | 50
days | 5.1 (2.4) | 6.1 (3.3)

3. Secondary Outcome: Number of Participants Who Were Readmitted to the Hospital
Description: Whether or not a patient was readmitted to the hospital within 30 days after the operation will be determined through chart review, clinical encounters, and phone calls.
Time Frame: 30 days post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Povidone-iodine Irrigation | No Irrigation
Number analyzed (Participants) | 50 | 50
Participants | 0 | 3

4. Secondary Outcome: Number of Participants Who Visited the Emergency Room
Description: Whether or not a patient visited the emergency room for care directly related to the operation within 30 days after the operation will be determined through chart review, clinical encounters, and phone calls.
Time Frame: 30 days post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Povidone-iodine Irrigation | No Irrigation
Number analyzed (Participants) | 50 | 50
Participants | 3 | 7

ADVERSE EVENTS:
Time Frame: 30 days post surgery
Arm/Group | Povidone-iodine Irrigation | No Irrigation
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-29): https://cdn.clinicaltrials.gov/large-docs/20/NCT02664220/Prot_SAP_000.pdf